CLINICAL TRIAL: NCT05004311
Title: An Open-label, Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Cenerimod After Single-dose Administration in Subjects With Severe Renal Impairment and Control Subjects
Brief Title: The Effect of Severe Kidney Impairment on Cenerimod Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID-064-107; 2021-001522-21 (EudraCT Number)
Record Dates: First submitted 2021-08-03; First posted 2021-08-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-08

CONDITIONS: Healthy; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — cenerimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (severe renal function impairment) (Experimental): Eight (8) participants with severe renal impairment.
  Interventions: Drug: Cenerimod
- Group B (healthy) (Experimental): Eight (8) control participants, matched to the 8 severe renal impaired participants enrolled in Group A.
  Interventions: Drug: Cenerimod

INTERVENTIONS:
Drug: Cenerimod — A single oral dose of 0.5 mg cenerimod will be administered as a film-coated tablet in the morning of Day 1 under fasted conditions
  Other Names: ACT-334441

SUMMARY:
To investigate the PK of cenerimod in participants with severe renal impairment as compared to healthy control participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Women of childbearing potential must have a negative serum pregnancy test at screening, a negative urine pregnancy test on Day -1, and agree to consistently and correctly use a highly effective method of contraception.
* Women of non-childbearing potential.
* Body mass index of 18.0 to 35.0 kg/m2 (inclusive) at Screening
* Negative SARS-CoV-2 reverse transcription polymerase chain reaction test on Day -1.

Additional inclusion criteria for participants with severe renal impairment

* Estimated glomerular filtration rate (eGFR) at screening using the Modification of Diet in Renal Disease formula less-than 30 mL/min/1.73 m2 for participants with renal impairment. The eGFR value should be confirmed on Day -1.
* Systolic blood pressure (SBP) 100 to 180 mmHg, diastolic BP (DBP) 50 to 105 mmHg, and pulse rate 60 to 100 bpm (inclusive), on Day 1 pre-dose.
* Stable concomitant medications for at least 3 weeks prior to screening and up to Day 1.
* Aspartate aminotransferase and alanine aminotransferase above the upper limit of normal.
* Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinanalysis) except for those related to renal impairment at Screening and on Day-1.

Additional inclusion criteria for control participants

* eGFR at Screening using the Modification of Diet in Renal Disease formula of ≥ 90 mL/min/1.73 m2.
* SBP 90 to 139 mmHg, DBP 60 to 89 mmHg, and pulse rate 60 to 99 bpm, measured on the same arm, after 5 min in the supine position at screening and on Day 1 pre-dose.

Exclusion Criteria:

* Pregnant or lactating women.
* Participation in a clinical study involving study treatment administration within 3 months prior to screening or participation in more than 2 clinical studies within 1 year prior to Screening.
* Previous exposure to cenerimod.
* Known hypersensitivity to any excipients of the treatment formulation.
* Clinically relevant abnormalities on a 12-lead electrocardiogram at Screening and Day -1.
* Previous treatment with anti-arrhythmic medications of class Ia or III within 2 weeks or 5 half-lives, whichever is longer, prior to study treatment administration.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study treatment except for renal disease, appendectomy, herniotomy, or cholecystectomy.
* Aspartate aminotransferase and alanine aminotransferase above the upper limit of normal.
* Legal incapacity or limited legal capacity at Screening.

Additional exclusion criteria for participants with severe renal impairment:

* Presence of severe cardiac disease.
* End-stage renal disease that requires dialysis.
* History of severe renal artery stenosis.
* Serum potassium concentration > 5.5 mmol/L.
* Presence of unstable diabetes mellitus.
* Strict fluid restriction.
* Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis) except for those related to renal impairment at Screening and on Day -1.

Additional exclusion criteria for control participants

* Clinically relevant findings on the physical examination at Screening.
* Clinically relevant findings in clinical laboratory tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t) of cenerimod | Total duration: up to 52 days
Area under the plasma concentration-time curve (AUC from 0 to infinity) of cenerimod | Total duration: up to 52 days
The maximum plasma concentration (Cmax) of cenerimod | Total duration: up to 52 days
The time to reach Cmax (tmax) of cenerimod | Total duration: up to 52 days
Terminal half-life (t½) of cenerimod | Total duration: up to 52 days
Apparent oral clearance (CL/F) of cenerimod | Total duration: up to 52 days
Extent of cenerimod protein plasma binding (PPB) | Total duration: up to 52 days
Apparent volume of distribution (Vz/F) of cenerimod | Total duration: up to 52 days

SECONDARY OUTCOMES:
Total lymphocyte count count. | Total duration: up to 66 days
Change from baseline at each time point of measurement in electrocardiogram QT interval | Total duration: up to 66 days
Change from baseline in body weight | Total duration: up to 66 days
Change from baseline in systolic and diastolic blood pressure (in the supine position) | Total duration: up to 66 days
Incidence of abnormal laboratory test results | Total duration: up to 66 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- BlueClinical Phase 1 Hospital de Prelado, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No